CLINICAL TRIAL: NCT06669065
Title: Assessment Of Scanning Accuracy of Maxillary Full-Arch Dental Implants Using Extraoral Vs Intraoral Scanning Techniques. [A Clinical Study]
Brief Title: Comparing Scanning Accuracy of Full-Arch Maxillary Implants: Extraoral vs. Intraoral Techniques
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Misr University for Science and Technology (Other)
Responsible Party: Principal Investigator, HEBA ELSARRIF, Principal Investigator, Lecturer of Removable Prosthodontics, Misr University for Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2024/0016
Record Dates: First submitted 2024-10-24; First posted 2024-11-01 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Edentulous Maxilla
Keywords: scanning of all on x maxillary dental implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- patients rehabilitated with dental implants in upper edentulous jaws (Experimental): patients rehabilitated with dental implants in upper edentulous jaws, then different data acquisition techniques will be applied to the patients using conventional impressions versus intra-oral scanning methods
  Interventions: Device: extraoral versus intraoral scanning techniques

INTERVENTIONS:
Device: extraoral versus intraoral scanning techniques — different data acquisition techniques for full-arch dental implants

SUMMARY:
Data acquisition from the patients:

After 4 months of implant placement, three impressions/scans will be made for each patient as follows:

Data 1: conventional impression using open tray transfer copings and silicon impression material. After cast verification, the scan bodies will be connected to the analogues on the master cast, which will be scanned using a laboratory scanner. The STL file will be used as a reference scan.

Data 2: The scan bodies will be connected to the implants intraorally, and an intraoral scan will be made using the intraoral scanner. The STL file will be stored for comparison.

Data 3: the scan bodies will be splinted using dental floss after being connected to the implants intraorally and then a scan will be made using the intraoral scanner. The STL file will be stored for comparison.

- Data alignment and accuracy measurements: The accuracy measurement will be done based on ISO 5725 in which a combination of trueness and precision was approved to define the accuracy of the measurement method. (15) The scanned data will be compared as follows: the STL files from the intraoral digital scans (data 2 and 3) and the extraoral scan of the master cast (data 1) will be imported into a 3D inspection software program that is a metrology program used to analyse and compare 3D meshes. The information for both reference and targets (the scanned data to be compared) will be uploaded into the program and the area of interest of 3D meshes will be marked, The "3D Compare" function will be employed by projecting all paired points with a colour-coded map created to display the deviation patterns of the investigated surfaces. The superimpositions will be used to assess the 3D accuracy for both the digital intraoral scans with the extraoral scan of the verified stone casts.

- Statistical analysis: Data will be collected, analysed, and then tabulated.

DETAILED DESCRIPTION:
Data acquisition from the patients:

After the osseointegration period of the dental implants, three impressions/scans will be made for each patient as follows:

1. Data #1: A conventional impression using open tray transfer copings will be connected to the dental implants intraorally and splinted together using dental floss and a duralay resin pattern to ensure complete fixation and immobility. Then, a custom acrylic resin tray with an open window and silicon impression material will be used for the final impression making. a master cast will be poured, and the transfer copings will be reconnected onto the implant analogues inside the cast to replicate implant positions intraorally. the transfer copings/impression posts will be connected with duralay resin pattern to form a verification jig assembly. The verification jig assembly will be connected to the implants inside the patient's mouth to check passivity, in case of improper passivity, the jig will be sectioned at areas between the implants and then reconnected with duraly and an impression will be repeated, if passivity is ensured, the verification jig assembly will be reconnected to the master cast that will be then deemed as a verified master cast. The next step after master cast verification is the connection of the scan bodies to the implant analogues then scanning it with a laboratory scanner to gain an STL file of the (control) group or the (reference) group of the research.
2. Data #2: The scan bodies will be connected to the implants intraorally, and an intraoral scan will be made using the intraoral scanner. The STL file will be stored for comparison. (comparator 1)
3. Data #3: scan bodies will be splinted together using dental floss and composite resin will be added to the floss at areas found between the scan bodies to add some irregularities, then a scan will be made using the intraoral scanner. The STL file will be stored for comparison. (comparator 2)

   * Data alignment and accuracy measurements:

The accuracy measurement will be done based on ISO 5725 in which a combination of trueness and precision was approved to define the accuracy of the measurement method. (15) The scanned data will be compared as follows: the STL files from the intraoral digital scans (data 2 and 3) and the extraoral scan of the master cast (data 1) will be imported into a 3D inspection software program that is a metrology program used to analyse and compare 3D meshes. The information for both reference and targets (the scanned data to be compared) will be uploaded into the program and the area of interest of 3D meshes will be marked, The "3D Compare" function will be employed by projecting all paired points with a colour-coded map created to display the deviation patterns of the investigated surfaces. The superimpositions will be used to assess the 3D accuracy for both the digital intraoral scans with the extraoral scan of the verified stone casts.

* Statistical analysis:
* Handling of numerical/quantitative variables:

Numerical data will be explored for normality by checking the data distribution using Kolmogorov- Smirnov and Shapiro-Wilk tests. Data will be presented as mean & standard deviation. If data will be normally distributed comparison between 2 different groups will be performed by using Independent t-test, a comparison between 2 related groups will be performed by using a Paired t-test, while a comparison between more than 2 groups will be performed by using A Way ANOVA test followed by Tukey's Post Hoc test for multiple comparisons.

If data will be non-parametric data comparison between 2 different groups will be performed by using the Mann-Whitney test, a comparison between 2 related groups will be performed by using the Wilcoxon Signed Rank test, while a comparison between more than 2 groups will be performed by using Kruskal-Wallis test.

- Handling of categorial/qualitative variables: Data will be presented as frequency and percentages. All comparisons will be performed by using the Chi-square test.

Statistical analysis:

Data will be collected, tabulated, and statistically analyzed using Microsoft Excel ® 2016, Statistical Package for Social Science (SPSS)® Ver. 24. and Minitab ® statistical software Ver. 16.

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous patients who had been wearing complete dentures and received 4 implants in the upper jaw.
2. Patients with no systemic diseases affecting bone remodelling and osseointegration.
3. Ridges showing well-keratinized mucosa.

Exclusion Criteria:

1. Smokers.
2. Non-compliant patients.
3. Patients with systemic diseases that may affect bone remodelling and osseointegration.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
assessment of accuracy of different intra oral scanning techniques versus the extraoral scanning method | 6 - 9 months
  The primary outcome of this study is to evaluate and compare the accuracy of various intraoral scanning techniques against a benchmark established by an extraoral scanning method. Accuracy will be measured using parameters such as dimensional precision, surface detail reproduction, and alignment with reference models. The study aims to determine which intraoral scanning technique provides results that are statistically comparable to or exceed the accuracy of the extraoral method, thereby informing best practices in dental imaging.

CONTACTS AND LOCATIONS:
Overall Officials: HEBA ELSARRIF, Principal Investigator — Misr University for Science and Technology
Locations (1):
- Misr University for Science and Technology, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, CSR
Time Frame: April 2025
Access Criteria: practitioners interested in the same field of research
URL: https://clinicaltrials.gov